CLINICAL TRIAL: NCT01069471
Title: Safety and Reactogenicity of a Candidate Vaccine Against S. Dysenteriae When Administered to Healthy Adults
Brief Title: Safety and Reactogenicity of Bioconjugate Vaccine to Prevent Shigella
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoVaxyn AG (Industry)
Responsible Party: Veronica Gambillara, GlycoVaxyn AG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SD 133
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Shigellosis
Keywords: S.dysenteriae; Healthy volunteers; Conjugate vaccine; Safety; Immunogenicity; Dose scaling
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Shigella Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HHD O1-EPA plus adjuvant (Experimental): 10 ug of Shigella dysenteriae polysaccharide O1 conjugated to EPA adjuvanted to aluminium hydroxide
  Interventions: Biological: Shigella vaccine
- HHD O1-EPA (Experimental): 10 ug of Shigella dysenteriae polysaccharide O1 conjugated to EPA
  Interventions: Biological: Shigella vaccine
- LHD O1-EPA adjuvanted (Experimental): 2 ug of Shigella dysenteriae polysaccharide O1 conjugated to EPA adjuvanted to aluminium hydroxide
  Interventions: Biological: Shigella vaccine
- LHD O1-EPA (Experimental): 2 ug of Shigella dysenteriae polysaccharide O1 conjugated to EPA
  Interventions: Biological: Shigella vaccine

INTERVENTIONS:
Biological: Shigella vaccine — Two intramuscular injections of bioconjugate vaccine will be administrated at D0 and D60.

SUMMARY:
Healthy volunteers will receive a 2-dose vaccination with Shigella dysenteriae candidate vaccine spaced 8 weeks apart. The objective is to demonstrate the safety and reactogenicity of the Shigella dysenteriae bioconjugate vaccine (GVXN SD133) alone or in combination with an adjuvant (Aluminium Hydroxide). The safety and reactogenicity of the GVXN SD133 vaccine will be also evaluated at two different concentrations of antigen, Shigella polysaccharide O1. Blood samples will be collected at intervals to examine systemic vaccine antigen-specific immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, aged between 18 and 50 years.
* Subjects who have undergone a detailed medical history, clinical checkup and are in good health.
* Subjects who have understood the purpose of the study and have freely signed the informed consent.
* Subjects who consent with repeated blood samples taking.
* Subjects who will be available to perform the follow-up visits, are reachable by telephone, and are able to complete the diary cards throughout the study duration.
* For female volunteers, a negative pregnancy test and an adequate contraception throughout the study duration.

Exclusion Criteria:

* Known history of recent contact Shigella infection or long-term residence in a Shigella endemic region (Central America, Africa, and India).
* Known history of hypersensitivity to any component of the vaccine (EPA; Aluminium Hydroxide).
* Subjects with compromised immune system.
* Family history of congenital or hereditary immunodeficiency.
* Chronic administration of an immunosuppressive treatment or other immune-modifying drugs within six months prior to the first vaccine dose.
* Subjects that received any other vaccine during the 1 month preceding the 1st injection and may receive before the 2nd injection. If the subject needs to be vaccinated during this period, he/she will be withdrawn from the study.
* Subjects suffering of a disease at the time of enrolment. 'Disease' is defined as the presence of a mild or severe illness with or without fever.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Any laboratory data collected during the screening phase found to be outside the normal range defined by the laboratory.
* Positive test for HIV, and evidence of HBV or HCV.
* Pregnant or breast-feeding women.
* History of alcohol, drug or psychotropic drug abuse (which interferes with a normal lifestyle) during the previous year.
* Subjects for which follow-up is compromised due to socio-cultural, geographic or psychological reasons.
* Any other significant finding that in the opinion of the Investigator that would increase the risk of having an adverse outcome from participating in the study.
* Subjects that are participating or have participated in another clinical trial in the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity of the bioconjugate vaccine, GVXN SD133 | Each study visits and at the and of the study

SECONDARY OUTCOMES:
Humoral immunogenicity | at day 0, 30, 60, 90 and 150

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hatz, Prof. Dr., Principal Investigator — Institute of Social and Preventive Medicine
Locations (1):
- Institute of Social and Preventive Medicine, Zurich, Switzerland

REFERENCES:
- [Derived] Hatz CF, Bally B, Rohrer S, Steffen R, Kramme S, Siegrist CA, Wacker M, Alaimo C, Fonck VG. Safety and immunogenicity of a candidate bioconjugate vaccine against Shigella dysenteriae type 1 administered to healthy adults: A single blind, partially randomized Phase I study. Vaccine. 2015 Aug 26;33(36):4594-601. doi: 10.1016/j.vaccine.2015.06.102. Epub 2015 Jul 7. PMID 26162850